CLINICAL TRIAL: NCT05056571
Title: The Effects of Online Progressive Muscle Relaxation Exercise on Occupational Stress, Headache and Well-being in Intensive Care Nurses
Brief Title: Progressive Muscle Relaxation Exercise on Intensive Care Nurses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Merve Gulbahar, Research Asisstant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E2-21-814
Record Dates: First submitted 2021-09-20; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Occupational Stress
Keywords: headache; intensive care units; occupational Stress; relaxation; well-being
MeSH Terms: conditions — Occupational Stress; Headache | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxation exercise (Experimental): Intensive care nurses will apply 20 minutes of online (zoom meeting) progressive muscle relaxation exercise twice a week, for 8 weeks, for a total of 16 group sessions. In order to support nurses' adaptation to the research, the group counselor will remind the nurses by phone twice a week during the implementation process, and their regular participation in online sessions will be supported.
  Interventions: Behavioral: Progressive muscle relaxation
- Control (No Intervention): No attempt will be made during the research.

INTERVENTIONS:
Behavioral: Progressive muscle relaxation — Progressive muscle relaxation exercise is a type of exercise in which tense muscles in your body gradually relax and relax. It is an application that allows you to forcefully stretch every muscle group in your body, hold it tight for 5 seconds, and then relax it. Visualize your tense muscles throughout this exercise and imagine that the feeling of relaxation spreads to all your muscles in the form of a wave and the tension is relieved. Keep breathing throughout the entire exercise.
  Arms: Relaxation exercise

SUMMARY:
Nurses who intensive care unit will be entered. Participants will be randomized to one of two study arms:

Arm 1: Progressive muscle relaxation; Arm 2: control. Hypothesis: Progressive muscle relaxation will decrease occupational stress, headache and improve well-being.

DETAILED DESCRIPTION:
Previous reports have revealed that non-pharmacological approaches such as aromatherapy, massage, meditation, music therapy, breathing exercises, yoga and progressive muscle relaxation exercises (PGE) have been used to reduce stress and fatigue of individuals and improve their well-being.

However, there have been limited studies that directly focus on supporting intensive care nurses who face serious problems with intense work tempo, experience excessive stress, headache, tension, fatigue, are open to psychosocial problems such as anxiety, depression and burnout.

Besides, till date, no study has been conducted to determine the effects of progressive relaxation exercise on occupational stress, headache and well-being for intensive care nurses.

The present study investigates the effects of progressive muscle relaxation in a single-site, 2-arm, assessor-blinded randomized, controlled study of 100 intensive care nurses.

Arm 1: relaxation; Arm 2: Attention matched control. The investigators hypothesize that progressive muscle relaxation will decrease the severity of occupational stress and headache and improve well-being.

ELIGIBILITY:
Inclusion Criteria:

* Working in cardiovascular intensive care for at least 6 months
* Having a headache at least once a week
* No physical disability
* Those who do not have a neurological diagnosis (having cerebrovascular disease, multiple sclerosis, etc.)
* No psychiatric diagnosis
* Not applying any complementary methods at the time the research was conducted.
* Nurses who volunteered to participate in the study

Exclusion Criteria:

* Nurses followed up with the diagnosis of end-stage renal disease, Chronic Obstructive Pulmonary Disease, advanced heart failure, chronic liver disease, musculoskeletal problem, hypothyroidism and depression
* Having physical and mental health problems that prevent communication
* Nurses who practiced any complementary method (relaxation exercise, yoga, etc.) during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Occupational Stress | Baseline measurements, at the end of 4., 8th week and one week after the completion of the interventions
  Occupational stress severity will be measured based on patient report by the Occupational Stress Scale.
  Higher scores indicate increased occupational stress.

SECONDARY OUTCOMES:
Change in headache severity | Baseline measurements, at the end of 4., 8th week and one week after the completion of the interventions
  Headache severity will be measured based on patient report by the Visual Analog Scale. Lower scores indicate low level of headache.
Change in Well-being | Baseline measurements, at the end of 4., 8th week and one week after the completion of the interventions
  Well-being will be measured by the Flourishing Scale. Higher scores on the scale mean better well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra G Metin, PhD, Principal Investigator — Hacettepe University Faculty of Nursing
Locations (1):
- Ankara City Hospital Cardiovascular Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No